CLINICAL TRIAL: NCT02388347
Title: A Phase 1a, Randomised, Placebo-controlled, Single-ascending Dose Study to Evaluate the Safety and Tolerability of MEDI7836 in Healthy Adults
Brief Title: A Study to Assess the Safety of MEDI7836 in Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5450C00001
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Participants will receive a single-dose of Placebo subcutaneous (SC) injection on Day 1.
  Interventions: Drug: Placebo SC
- MEDI7836 Dose 1 (Experimental): Participants will receive a single-dose of MEDI7836 Dose 1 SC injection on Day 1.
  Interventions: Biological: MEDI7836 Dose 1
- MEDI7836 Dose 2 (Experimental): Participants will receive a single-dose of MEDI7836 Dose 2 SC injection on Day 1.
  Interventions: Biological: MEDI7836 Dose 2
- MEDI7836 Dose 3 (Experimental): Participants will receive a single-dose of MEDI7836 Dose 3 SC injection on Day 1.
  Interventions: Biological: MEDI7836 Dose 3
- MEDI7836 Dose 4 (Experimental): Participants will receive a single-dose of MEDI7836 Dose 4 SC injection on Day 1.
  Interventions: Biological: MEDI7836 Dose 4

INTERVENTIONS:
Drug: Placebo SC — Participants will receive a single-dose of Placebo subcutaneous (SC) injection on Day 1.
  Arms: Placebo
Biological: MEDI7836 Dose 1 — Participants will receive a single-dose of MEDI7836 Dose 1 SC injection on Day 1.
  Arms: MEDI7836 Dose 1
Biological: MEDI7836 Dose 2 — Participants will receive a single-dose of MEDI7836 Dose 2 SC injection on Day 1.
  Arms: MEDI7836 Dose 2
Biological: MEDI7836 Dose 3 — Participants will receive a single-dose of MEDI7836 Dose 3 SC injection on Day 1.
  Arms: MEDI7836 Dose 3
Biological: MEDI7836 Dose 4 — Participants will receive a single-dose of MEDI7836 Dose 4 SC injection on Day 1.
  Arms: MEDI7836 Dose 4

SUMMARY:
To assess the safety of a single ascending dose of MEDI7836 in healthy adult male subjects and healthy adult female subjects of non-childbearing potential.

DETAILED DESCRIPTION:
This is a Phase 1a, randomised, blinded (the investigator and subject will be blinded to treatment assignment and sponsor will be unblinded to treatment assignment), placebo-controlled study to evaluate the safety of single-ascending SC doses of MEDI7836 in healthy adult males subjects and healthy adult female subjects of non-childbearing potential. The study will be conducted at a single site in the United Kingdom (UK). Four dosing cohorts of MEDI7836 or placebo are planned for this study for a total of 32 subjects (24 subjects receiving MEDI7836, 8 subjects receiving placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Vital signs, ECG, and laboratory parameters within normal range at screening and Day -1
2. Negative alcohol and drug screen at screening and Day -1
3. Able and willing to comply with the requirements of the protocol
4. Females subjects must have been surgically sterilised or be postmenopausal
5. Nonsterilised males who are sexually active with a female partner of childbearing potential or a female partner who has been surgically sterilised by bilateral tubal ligation must use a condom with spermicide with their partner from screening until the end of the study follow-up period

Exclusion Criteria:

1. Concurrent enrolment in another clinical study where the subject is receiving an investigational product
2. Individuals who are legally institutionalised
3. Receipt of any marketed or investigational biologic agent within 4 months
4. Receipt of any investigational non-biologic agent within 3 months or 5 half-lives prior to screening, whichever is longer
5. Use of any medication (prescription or over the counter, including herbal remedies) within 14 days or 5 half-lives of Day 1,
6. Known history of allergy or reaction to any component of the investigational product formulation
7. History of anaphylaxis following any biologic therapy
8. History of chronic alcohol or drug abuse within 12 months prior to screening,
9. Presence of a positive drug or alcohol screen at screening and Day -1.
10. Current smoker, or history of smoking within 6 months of screening
11. Pregnant or breastfeeding women
12. Any active medical or psychiatric condition or other reason which, in the opinion of the investigator or medical monitor, may compromise the safety of the subject in the study or interfere with evaluation of the investigational product or reduce the subject's ability to participate in the study
13. Any clinically relevant abnormal findings in physical examination, ECG, vital signs, haematology, clinical chemistry or urinalysis during screening or Day -1,
14. History of any known primary immunodeficiency disorder or use of immunosuppressive medication within 12 months of screening
15. History of a clinically significant infection requiring antibiotics or antiviral medication from 30 days prior to screening, up to and including Day 1
16. Diagnosis of a helminth parasitic infection within 6 months prior to screening that has not been treated with, or has failed to respond to, standard of care therapy
17. History of cancer, except for basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success with curative therapy ≥ 12 months prior to screening or other malignancies treated with apparent success with curative therapy ≥ 5 years prior to screening
18. Positive tuberculosis (TB) test (Quantiferon-TB Gold) at screening or TB requiring treatment within the 12 months prior to the screening visit
19. Positive hepatitis B surface antigen, hepatitis B anti-core antibody, or hepatitis C virus antibody serology at screening.
20. Subjects with a history of hepatitis B vaccination without history of hepatitis B are allowed to enter the study.
21. A positive human immunodeficiency virus test at screening or subject taking antiretroviral medications, as determined by medical history and/or subject's verbal report
22. Evidence of active liver disease, including jaundice or aspartate transaminase (AST), alanine transaminase (ALT), or alkaline phosphatase greater than twice the upper limit of normal (ULN)
23. Major surgery within 8 weeks prior to screening, or planed in-patient surgery or hospitalisation during the study period
24. Receipt of live attenuated vaccines 30 days prior to the date of screening Where participation in the study would result in donation of blood or blood products in excess of 500 mL within an 8-week period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annelize Koch, MD, Principal Investigator — Parexel
Locations (1):
- Research Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 79 participants were screened. Of these, 32 participants were randomized and treated in the study.
Groups:
- Placebo: Participants received a single-dose of Placebo subcutaneous (SC) injection on Day 1.
- MEDI7836 Dose 1: Participants received a single-dose of MEDI7836 Dose 1 subcutaneous (SC) injection on Day 1.
- MEDI7836 Dose 2: Participants received a single-dose of MEDI7836 Dose 2 subcutaneous (SC) injection on Day 1.
- MEDI7836 Dose 3: Participants received a single-dose of MEDI7836 Dose 3 subcutaneous (SC) injection on Day 1.
- MEDI7836 Dose 4: Participants received a single-dose of MEDI7836 Dose 4 subcutaneous (SC) injection on Day 1.
Period: Overall Study
Arm/Group | Placebo | MEDI7836 Dose 1 | MEDI7836 Dose 2 | MEDI7836 Dose 3 | MEDI7836 Dose 4
Started | 8 | 6 | 6 | 6 | 6
Completed | 8 | 6 | 5 | 6 | 6
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: As Treated Population included all randomized participants and treated with MEDI7836 or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI7836 Dose 1 | MEDI7836 Dose 2 | MEDI7836 Dose 3 | MEDI7836 Dose 4 | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.4 (9.9) | 38.2 (7.1) | 32.8 (11.5) | 32.8 (9.7) | 32.0 (14.0) | 34.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 6 | 6 | 6 | 6 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment- Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: Any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening situation (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of a participant who received MEDI7836. Treatment-emergent adverse events between administration of investigational product and Day 281 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From Study Drug Administration to 281 Days Postdose
Population: As Treated Population included all randomized participants and treated with MEDI7836 or placebo.
Measure: Number; unit: Participant
Arm/Group | Placebo | MEDI7836 Dose 1 | MEDI7836 Dose 2 | MEDI7836 Dose 3 | MEDI7836 Dose 4
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Participant
  TEAEs | 6 | 4 | 6 | 5 | 6
  TESAEs | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Injection Site Reactions
Description: Participants were evaluated for manifestations of injection site reactions.
Time Frame: From Study Drug Administration to 281 Days Postdose
Population: As Treated Population included all randomized participants and treated with MEDI7836 or placebo.
Measure: Number; unit: Participant
Arm/Group | Placebo | MEDI7836 Dose 1 | MEDI7836 Dose 2 | MEDI7836 Dose 3 | MEDI7836 Dose 4
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Participant | 4 | 2 | 3 | 0 | 5

3. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as Treatment-Emergent Adverse Events
Description: An abnormal laboratory finding which required an action or intervention by the investigator, or a finding judged by the investigator to represent a change beyond the range of normal physiologic fluctuation were reported as an adverse event. Treatment-emergent adverse events between first dose of study drug and Day 281 after the last dose that were absent before treatment or that worsened relative to pre-treatment state. Laboratory evaluations (haematology, serum chemistry and urinalysis) of blood and urine samples were performed.
Time Frame: From Study Drug Administration to 281 Days Postdose
Population: As Treated Population included all randomized participants and treated with MEDI7836 or placebo.
Measure: Number; unit: Participant
Arm/Group | Placebo | MEDI7836 Dose 1 | MEDI7836 Dose 2 | MEDI7836 Dose 3 | MEDI7836 Dose 4
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Participant
  Platelet count decreased | 0 | 1 | 0 | 0 | 0
  Aspartate aminotransferase increased | 0 | 0 | 0 | 1 | 1
  Transaminases increased | 1 | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Vital Signs and Physical Examination Abnormalities Reported as Treatment-Emergent Adverse Events
Description: Vital sign parameters included blood pressure, temperature, pulse rate, respiratory rate and weight. Physical examination included assessment of general appearance, weight, head, ears, eyes, nose, throat, neck, skin, cardiovascular system, respiratory system, abdominal system, and nervous system. Criteria for abnormal physical findings was based on investigator's discretion. TEAEs were present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug until Day 281 after the last dose of study drug.
Time Frame: From Study Drug Administration to 281 Days Postdose
Population: As Treated Population included all randomized participants and treated with MEDI7836 or placebo.
Measure: Number; unit: Participant
Arm/Group | Placebo | MEDI7836 Dose 1 | MEDI7836 Dose 2 | MEDI7836 Dose 3 | MEDI7836 Dose 4
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Participant | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities Reported as Treatment-Emergent Adverse Events
Description: AEs observed in participants with clinically significant ECG abnormalities were assessed. ECG parameters included heart rate, RR, PR, QRS, QT and QTc intervals. Treatment-emergent adverse events between administration of investigational product and Day 281 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: From Study Drug Administration to 281 Days Postdose
Population: As Treated Population included all randomized participants and treated with MEDI7836 or placebo.
Measure: Number; unit: Participant
Arm/Group | Placebo | MEDI7836 Dose 1 | MEDI7836 Dose 2 | MEDI7836 Dose 3 | MEDI7836 Dose 4
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Participant | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Area Under the Concentration-Time Curve From Zero to Infinity (AUC [0-infinity]) of MEDI7836
Description: Area under the concentration-time curve of the MEDI7836 in serum over the time interval from 0 extrapolated to infinity (AUC0-inf).
Time Frame: Predose on Day 1 and on Days 2, 3, 4, 6, 8, 10, 15, 29, 43, 57, 85, 113, 169, 225 and 281 Postdose
Population: Pharmacokinetic (PK) Population included all participants who received MEDI7836 had detectable postdose MEDI7836 serum concentrations.
Measure: Mean (Standard Deviation); unit: Day*microgram per milliliter
Arm/Group | MEDI7836 Dose 1 | MEDI7836 Dose 2 | MEDI7836 Dose 3 | MEDI7836 Dose 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
Day*microgram per milliliter | 62.958 (29.629) | 310.805 (204.858) | 807.725 (418.083) | 1101.742 (817.295)

7. Secondary Outcome: Area Under the Concentration-Time Curve From Zero to Last Observation (AUC [0-t]) of MEDI7836
Description: Area under the concentration-time curve of the MEDI7836 in serum over the time interval from 0 to the last quantifiable data point (AUC0-t).
Time Frame: Predose on Day 1 and on Days 2, 3, 4, 6, 8, 10, 15, 29, 43, 57, 85, 113, 169, 225 and 281 Postdose
Population: PK Population included all participants who received MEDI7836 had detectable postdose MEDI7836 serum concentrations.
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | MEDI7836 Dose 1 | MEDI7836 Dose 2 | MEDI7836 Dose 3 | MEDI7836 Dose 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
day*mcg/mL | 62.106 (29.237) | 308.965 (203.367) | 799.769 (406.585) | 1096.620 (807.266)

8. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of MEDI7836
Description: The Cmax is the maximum observed serum concentration of study drug.
Time Frame: Predose on Day 1 and on Days 2, 3, 4, 6, 8, 10, 15, 29, 43, 57, 85, 113, 169, 225 and 281 Postdose
Population: PK Population included all participants who received MEDI7836 had detectable postdose MEDI7836 serum concentrations.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | MEDI7836 Dose 1 | MEDI7836 Dose 2 | MEDI7836 Dose 3 | MEDI7836 Dose 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
microgram per milliliter (mcg/mL) | 1.587 (0.436) | 10.435 (1.520) | 24.600 (5.313) | 41.933 (7.208)

9. Secondary Outcome: Apparent Systemic Clearance (CL/F) of MEDI7836
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: Predose on Day 1 and on Days 2, 3, 4, 6, 8, 10, 15, 29, 43, 57, 85, 113, 169, 225 and 281 Postdose
Population: PK Population included all participants who received MEDI7836 had detectable postdose MEDI7836 serum concentrations.
Measure: Mean (Standard Deviation); unit: milliliter per day (mL/day)
Arm/Group | MEDI7836 Dose 1 | MEDI7836 Dose 2 | MEDI7836 Dose 3 | MEDI7836 Dose 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
milliliter per day (mL/day) | 616.206 (422.587) | 481.219 (282.488) | 463.827 (226.960) | 706.952 (283.588)

10. Secondary Outcome: Terminal Phase Elimination Half Life (T1/2) of MEDI7836
Description: Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the serum.
Time Frame: Predose on Day 1 and on Days 2, 3, 4, 6, 8, 10, 15, 29, 43, 57, 85, 113, 169, 225 and 281 Postdose
Population: PK Population included all participants who received MEDI7836 had detectable postdose MEDI7836 serum concentrations.
Measure: Mean (Standard Deviation); unit: day
Arm/Group | MEDI7836 Dose 1 | MEDI7836 Dose 2 | MEDI7836 Dose 3 | MEDI7836 Dose 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
day | 26.988 (14.902) | 28.091 (14.121) | 36.944 (9.329) | 37.013 (5.185)

11. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of MEDI7836
Description: The Tmax is defined as actual sampling time to reach maximum observed MEDI7836 concentration.
Time Frame: Predose on Day 1 and on Days 2, 3, 4, 6, 8, 10, 15, 29, 43, 57, 85, 113, 169, 225 and 281 Postdose
Population: PK Population included all participants who received MEDI7836 had detectable postdose MEDI7836 serum concentrations.
Measure: Median (Full Range); unit: day
Arm/Group | MEDI7836 Dose 1 | MEDI7836 Dose 2 | MEDI7836 Dose 3 | MEDI7836 Dose 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
day | 4.0 [4 to 15] | 5.0 [3 to 8] | 5.0 [3 to 10] | 6.0 [4 to 10]

12. Secondary Outcome: Apparent Terminal-Phase Volume of Distribution (Vz/F) of MEDI7836
Description: The apparent volume of distribution of MEDI7836 after a single dose, calculated according to the equation: Vz/F = Apparent total clearance (CL/F) / terminal phase rate constant (λz).
Time Frame: Predose on Day 1 and on Days 2, 3, 4, 6, 8, 10, 15, 29, 43, 57, 85, 113, 169, 225 and 281 Postdose
Population: PK Population included all participants who received MEDI7836 had detectable postdose MEDI7836 serum concentrations.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MEDI7836 Dose 1 | MEDI7836 Dose 2 | MEDI7836 Dose 3 | MEDI7836 Dose 4
Number analyzed (Participants) | 6 | 6 | 6 | 6
mL | 18885.105 (7689.663) | 15032.685 (6066.111) | 22930.365 (8180.111) | 36686.872 (14142.345)

13. Secondary Outcome: Percentage of Participants Positive for Anti-Drug Antibodies to MEDI7836
Description: A participant was considered ADA-positive across the study if they had a positive reading at any time point during the study.
Time Frame: Predose on Day 1 to 281 days Postdose
Population: As Treated Population included all randomized participants and treated with MEDI7836 or placebo. Here, "n" is number of participants analysed at given time point.
Measure: Number; unit: Percentage of participant
Arm/Group | Placebo | MEDI7836 Dose 1 | MEDI7836 Dose 2 | MEDI7836 Dose 3 | MEDI7836 Dose 4
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Percentage of participant
  Baseline (n=8,6,6,6,6) | 25.0 | 33.3 | 66.7 | 50.0 | 50.0
  Post-Baseline Day 281 (n=8,6,5,6,6) | 12.5 | 66.7 | 20.0 | 50.0 | 50.0

ADVERSE EVENTS:
Time Frame: From Study Drug Administration to 281 Days Postdose
Arm/Group | Placebo | MEDI7836 Dose 1 | MEDI7836 Dose 2 | MEDI7836 Dose 3 | MEDI7836 Dose 4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/8 | 4/6 | 6/6 | 5/6 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | MEDI7836 Dose 1 (N=6) | MEDI7836 Dose 2 (N=6) | MEDI7836 Dose 3 (N=6) | MEDI7836 Dose 4 (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 4 (6) | 2 (2) | 3 (3) | 0 (0) | 5 (11)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (5) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.